CLINICAL TRIAL: NCT06180759
Title: Acute Analgesic Effects of DMT on Experimentally Induced Acute Nociceptive Pain, Hyperalgesia and Allodynia in Healthy Participants
Brief Title: Acute Analgesic Effects of DMT on Experimentally Induced Pain in Healthy Participants
Acronym: DPS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2023-01813
Record Dates: First submitted 2023-11-20; First posted 2023-12-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: On 3 separate days, participants will be administered DMT, ketamine or placebo in a randomized, counter-balanced order. Their effect on experimentally induced acute pain will be evaluated and compared.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous infusion of DMT (Experimental): Participants will be administered intravenous DMT.
  Interventions: Drug: Intravenous infusion of DMT
- Intravenous infusion of ketamine (Active Comparator): Participants will be administered intravenous racemic ketamine.
  Interventions: Drug: Intravenous infusion of ketamine
- Intravenous infusion of placebo (Placebo Comparator): Participants will be administered intravenous lacebo (saline infusion).
  Interventions: Drug: Intravenous infusion of placebo

INTERVENTIONS:
Drug: Intravenous infusion of DMT — A dose rate of 1.2 mg/min will be administered
  Arms: Intravenous infusion of DMT
Drug: Intravenous infusion of ketamine — A dose rate of 1.0 mg/min will be administered
  Arms: Intravenous infusion of ketamine
Drug: Intravenous infusion of placebo — A Placebo (saline infusion) will be administered.
  Arms: Intravenous infusion of placebo

SUMMARY:
N,N-dimethyltryptamine (DMT) is a classical psychedelic with similar effects like LSD or psilocybin. Preliminary evidence from case series and small open-label trials suggests that psychedelics may be promising candidates for the treatment of several pain-related diseases such as chronic pain, migraine, cluster headache or phantom limb pain. However, data from rigorously conducted and randomized clinical trials are lacking. Additionally, the potential acute analgesic properties of psychedelics remain poorly characterized. Therefore, the investigators will evaluate the efficacy of DMT on different pain qualities within a model of electrically induced pain in healthy participants. The analgesic effects will be compared to racemic ketamine (active control) and placebo within a cross-over design.

DETAILED DESCRIPTION:
Preliminary evidence from case series and small open-label trials suggests that psychedelics may be promising candidates for the treatment of several pain-related diseases such as chronic pain, migraine, cluster headache or phantom limb pain. However, data from rigorously conducted and randomized clinical trials are lacking. Additionally, the potential acute analgesic properties of psychedelics remain poorly characterized. For instance, it is unclear whether psychedelics possess acute antinociceptive effects or if they rather modulate secondary pain phenomena such as hyperalgesia, allodynia, and/or functional pain. Here, the investigators will employ a validated electrical stimulation model in healthy volunteers that produces acute nociceptive pain but also features of chronic pain such as hyperalgesia and allodynia. The model is established for the detailed assessment of the analgesic effect of known analgesics or new compounds. Thus, the investigators will evaluate the efficacy of N,N-dimethyltryptamine (DMT), a classical and naturally-occurring psychedelic, on different pain qualities within this model. DMT differs from other classical psychedelics in its very short elimination half-life. Due to its rapid metabolization by monoaminoxidases (MAO), DMT is not orally bioavailable in the absence of MAO-inhibitors and thus has to be administered continuously and intravenously. Recently, the investigators tested several continuous intravenous administration regimes of DMT that lead to the induction of a constant and rapidly adaptable psychedelic state. The regime allows to induce stable DMT effect that can be terminated rapidly. Due to this controllability, a continuous infusion of intravenous DMT is most suitable to assess time and concentration-dependent analgesic effects within the used pain model. The analgesic efficacy of DMT will be compared to ketamine, a known analgesic (positive control), and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 75 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study 6. Willing not to operate heavy machinery for 24 hours after the study session.

7. Willing to use effective birth control throughout study participation 8. Body mass index between 18-29 kg/m2 and body weight within 50 - 90kg

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic and/or dissociative substance use (not including cannabis) more than 15 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) scores (0 - 10) | During the infusion (55minutes)
  Difference of the cumulative NRS scores (area under the effect curves (AUECs)) between the DMT, ketamine (active-control) and placebo condition. NRS 0 represents "no pain at all" whereas 10 represents "the worst pain ever possible".

SECONDARY OUTCOMES:
Area of hyperalgesia and allodynia | During the electrical stimulation (2 hours)
  Difference of the cumulative areas of hyperalgesia and allodynia (Area under the effect curves (AUECs), in square centimeters * minutes) between the DMT, ketamine and placebo condition.
NRS scores after infusion | After stopping the infusion (65 minutes)
  Difference of the cumulative NRS scores (Area under the effect curves (AUECs)) between the DMT, ketamine and placebo condition
Association of subjective effect ratings with pain scores | During the electrical stimulation (2 hours)
  Assessment of the correlation between subjective effect ratings and NRS pain scores, areas of hyperalgesia and allodynia. Subjective effects are measured on the subjective effects scale (SES) that ranges from 0 ( = no effects) to 10 ( = most extreme effects).
Sensory and affective pain scores | Retrospective evaluation after the electrial stimulation at the end of each study session.
  Difference of retrospectively evaluated sensory and affective pain scores (Short version of the McGill Pain Questionnaire, SF-MPQ-D) between the DMT, ketamine and placebo condition. The SF-MPQ-D is scored from 0 (= no pain) to 3 (= strongest possible pain).
Association of psychedelic and mystical-type effects with pain scores | During the electrical stimulation (2 hours) and retrospective evaluation at the end of each study session.
  Correlation between psychedelic and mystical-type effects (Five Dimensional Altered states of consciousness (5D-ASC), States of Consciousness Questionnaire (SCQ)) with NRS pain scores and areas of hyperalgesia and allodynia.
Plasma levels of DMT and ketamine | During the electrical stimulation (2 hours)
  Plasma levels of DMT and ketamine over time
Association of the intensity of electrical currents with NRS pain scores | During the electrical stimulation (2 hours)
  Association of the intensity of electrical currents (in mA) that induced a target baseline pain score (NRS) of 6/10 with NRS pain scores and areas of hyperalgesia and allodynia.
Psychometric comparison between DMT, ketamine and placebo | During the electrical stimulation (2 hours) and retrospective evaluation at the end of each study session.
  Comparison of subjective effects, altered state of consciousness and mystical effect scores between DMT, ketamine, and placebo.
Effect modulation through personality traits | During the electrical stimulation (2 hours) and retrospective evaluation at the end of each study session.
  Effect modulation through personality traits (NEO-Five Factor Inventary (NEO-FFI), Saarbrücken Persönlichkeitsfragebogen (SPF), Elliots humility scale (EHS), Defense-style questionnaire-40 (DSQ-40), Connor-Davidson Resilience Scale (CD-RISC), Five Facet Mindfulness Scale (FFMQ), ABC Connectedness to Nature Scale, (ABC-CNS)).
Modulation of personality traits by acute subjective effects | During the electrical stimulation (2 hours) and retrospective evaluation at the end of each study session.
  Modulation of personality traits resilience (Connor-Davidson Resilience Scale, CD-RISC), mindfulness (Five Facet Mindfulness Questionnaire (FFMQ) and connectedness to nature (ABC-CNS) in association with acute subjective effects (Subjective Effects Scale (SES)) and psychedelic/mystical-type effects (Five Dimensional Altered States of consciousness Scale (5D-ASC), States of Consciousness Questionnaire (SCQ).
Autonomic effects | During the electrical stimulation (2 hours)
  Autonomic effects over time (blood pressure in mmHg, heart rate in beats per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland